CLINICAL TRIAL: NCT06742008
Title: DCM Anti-Heart Antibody Diagnostic Kit Study--assessment of the Predictive Value of Anti-beta1AR and Anti-L-CaC Antibodies in the Evolution to Dilated Cardiomyopathy in Patients With Acute Viral Myocarditis
Brief Title: Assessment of the Predictive Value of Anti-beta1AR and Anti-L-CaC Antibodies in the Evolution to Dilated Cardiomyopathy in Patients With Acute Viral Myocarditis
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: Jing yuan-VMC cohort study
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Viral Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples remaining after completion of routine clinical blood tests will be destroyed in accordance with the regulations of the hospitals in which the centers are located. The study doctor will take an additional 5ml of blood sample for AHA testing in addition to the routine clinical blood tests. Prior consent will be obtained from the patients before the blood samples are taken; after the completion of this study, the remaining blood samples from the additional 5 ml of blood samples will be approved by the Ethics Committee and will be used for future studies of DCM and the development of VMC in high-risk populations in accordance with ethical requirements.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background of the study Studies have shown that about one-third of patients with acute viral myocarditis (AVMC) eventually develop dilated cardiomyopathy (DCM), and that the autoimmune response to viral infection is key to the development of AVMC to DCM. A variety of antimyocardial autoantibodies (AHAs) are detected in the sera of patients with myocarditis. Among them, anti-β1AR antibodies are thought to contribute to the transition of AVMC to DCM possibly by promoting myocardial injury, cardiac remodeling, and impaired cardiac function. The role of anti-L-CaC antibodies in the evolution of AVMC to DCM is unknown, but they have been shown to induce ventricular tachycardia by increasing calcium inward flow and triggering early afterdepolarization, increasing the rate of sudden death and all-cause mortality in patients. Therefore, monitoring the levels of these antibodies may be useful in assessing the prognosis of patients with viral myocarditis. In this study, we propose to use a multicenter, prospective cohort study to further accurately assess the predictive value of these autoantibodies in the evolution of AVMC patients to DCM by detecting the serum levels of anti-β1AR antibodies and anti-L-CaC antibodies in AVMC patients and combining them with the clinical data and follow-up data, so as to provide prognostic biomarkers as well as targets for targeted interventions in AVMC.

Objective of the study A multicenter, prospective cohort study of the value of anti-β1AR and anti-L-CaC antibodies in the progression of AVMC patients to DCM, enrolling 300 AVMC patients, to further accurately assess the predictive value of anti-β1AR and anti-L-CaC antibodies in the progression of AVMC patients to DCM, and provide prognostic biomarkers and targeted interventions for AVMC. The study will provide prognostic biomarkers and targeted intervention for AVMC.

ELIGIBILITY:
Inclusion Criteria:

1. Meets diagnostic criteria for VMC
2. Clinical symptoms present for no more than 30 days
3. Age ≥ 18 years and ≤ 75 years
4. Subjects or their legal guardians are fully informed of the nature and risks of the study, participate voluntarily, and sign an informed consent form.

Exclusion Criteria:

1. Serious uncontrolled infection at enrolment ("uncontrolled" is defined as signs and symptoms of infection that persist without improvement despite antimicrobial or other treatment)
2. Uncontrolled active bleeding at enrollment
3. Systemic autoimmune disease such as systemic lupus erythematosus or diagnosed immunodeficiency disease at enrollment
4. Pregnancy or breastfeeding
5. Combination of serious diseases affecting survival, such as tumors, with a life expectancy shorter than 3 months
6. Patients with poor compliance who are unable to complete the full course of the study
7. Other conditions (e.g., overstimulation, sensitivity, cognitive impairment, mental illness, or substance abuse/addiction) that, in the judgment of the investigator, may increase the risk to the subject or interfere with the clinical study and judgment of the results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Viral myocarditis (VMC) is an inflammation of the myocardium caused by viral infections. Common viruses include coxsackievirus, adenovirus, cytomegalovirus, and influenza virus. The prognosis for patients with Acute viral myocarditis (AVMC) varies widely, with most patients recovering with treatment, but some progressing to dilated cardiomyopathy (DCM). Studies have shown that about one-third of patients with AVMC eventually develop DCM, and that the immune response following viral infection is key to the development of DCM in AVMC. Following viral infection, specific antigenic determinants within cardiomyocytes are exposed to the immune system, triggering an autoimmune response against the myocardium, leading to damage and dysfunction of cardiomyocytes.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of evolution to DCM in patients positive for anti-β1AR antibodies and anti-L-CaC antibodies | End of months 1, 3 and 6

SECONDARY OUTCOMES:
All-Cause Death, Rehospitalization for Heart Failure, or Sudden Death in Patients Positive for Anti-β1AR Antibodies and Anti-L-CaC Antibodies | End of months 1, 3 and 6

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, 430022, China, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No